CLINICAL TRIAL: NCT05197582
Title: The Effect of Tele-Health Application on Anxiety Level and Quality of Life of Patients in COVID-19 Quarantine: A Quasi-experimental Study
Brief Title: The Effect of Telemonitoring on Anxiety and Quality of Life in Patients in COVID 19 Quarantine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Arzu Bahar, assistant professor, Yuksek Ihtisas University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YuksekIU-ABAHAR-001
Record Dates: First submitted 2022-01-11; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pandemic
Keywords: telemedicine; anxiety; quarantine; Quality of Life
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A Clinical trial with experimental and control groups with
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-monitoring group (Active Comparator): The researchers called the patients in the experimental group on the first day of the quarantine and explained the topics covered in the COVID 19 patient education booklet to the patients. Patient education and follow-up in quarantine took approximately 25-30 minutes for each patient in the experimental group. The patients in quarantine were followed up by the researchers two more times, on the 5th and 9th days of the quarantine. On the 10th and last day of the quarantine, post-test online questionnaires were sent to the patients for the second time, and the data collection phase was ended.
  Interventions: Other: tele-monitoring
- Plasebo group (No Intervention): The patients in the control group were called by the researchers on the first day of the quarantine and asked to fill in the online pre-test forms. On the 10th day, the last day of the quarantine, the patients were called and the online post-test forms were sent for the second time, and the data were collected. There was no telephone follow up in the control group and the patients received only routine care in the home

INTERVENTIONS:
Other: tele-monitoring — The symptoms of the patients were evaluated by calling the patients on the 1st, 5th, and 9th days of the quarantine by the researchers.
  Arms: Tele-monitoring group

SUMMARY:
The study was carried out to evaluate the effect of telemonitoring service to be given to patients kept under quarantine during the COVID 19 pandemic on anxiety and quality of life.

DETAILED DESCRIPTION:
The COVID 19 pandemic, which continues today, has caused radical changes in social, cultural, education, and health systems around the world(Zhang and Liu 2020; Wang et all 2020; Alipour &Abdolahzadeh 2020). In this period, health care providers tried to use telehealth services as a good alternative to solve the problems caused by quarantine, social isolation practices to reduce the rate of transmission of the disease, and the limitation of physical access to health services due to the risk of transmission.

Thus, the use of telehealth applications, which first started in the 1950s, gained momentum especially during the pandemic period (Byrne 2020; Lurie & Carr 2018; Clipper 2020; Fagherazzi 2020). Telehealth applications, which have the opportunity to be widely used during the COVID 19 pandemic period, are generally a system that provides two-way communication between healthcare professionals and patients and includes image, speech, and digital communication technologies (Hazin & Qaddoumi, 2010; Merz et all 2021; Bryne 2020). Tele-monitoring is a good option to support patients in the management of existing physical symptoms of quarantined patients who are isolated at home, except for patients who need outpatient or hospital treatment in the COVID 19 pandemic. In studies investigating the presence of mental problems as a result of the decrease in the social support of the patients in this group due to social isolation, the study results indicate that the patients experience negative conditions such as depression, stress, sleep problems, and anxiety (Verma 2020, Alipour et all 2020; Chakeri et all 2020).

Therefore, when quarantined patients are evaluated holistically, there is a need for studies evaluating the effect of telehealth services to increase the quality of life by coping with mental problems such as anxiety and depression. Although there are studies in the related literature showing that telemonitoring can cope with physical problems, improve quality of life, and reduce mental problems such as anxiety and depression, studies showing the effect of telemonitoring given to quarantined patients on anxiety and quality of life are quite limited (Kamei et all 2021; Jahromi et all 2016; Charekei et all 2020; Allipour et all 2020). For this reason, our study was carried out to evaluate the effect of telemonitoring service to be given to patients kept under quarantine during the COVID 19 pandemic on anxiety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

- Volunteer patients who were diagnosed with COVID 19, over the age of 18, had no communication problems, were literate, had no diagnosed mental pathology, were able to use smartphones were included in the study

Exclusion Criteria:

* In the study, a patient whose general condition deteriorated during the COVID 19 quarantine and was hospitalized was excluded from the sample

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The MOS 36 Item Short Form Health Survey(SF-36) | 10 days after
  Scores of SF 36-Quality of Life Scale The scale consists of 8 subscales, including physical function, social function, physical role function, emotional role function, mental health, vitality, pain, and general health, and a total of 36 items. Evaluation in the scale is Likert type except for some items and the last 4 weeks are taken into consideration. Subscales evaluate health between 0-100 and the higher the score, the better the quality of life.

SECONDARY OUTCOMES:
The Beck Anxiety Scale | 10 days after
  The scores of the Beck Anxiety Scale It is a Likert-type assessment tool in which scores ranging from 0 to 3 are given in the 21-item scale. 8-15 points obtained from the scale = Mild anxiety, 16-25 points = Moderate anxiety, 26-63 points = Severe anxiety. While the lowest score that can be taken from the scale is 0, the highest score that can be obtained from the scale is 63. A high total score indicates an increase in anxiety severity

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Bahar, PhD, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Arzu Bahar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No